CLINICAL TRIAL: NCT01396616
Title: Clinical Evaluation of Toric Intraocular Lens Made by Aurolab
Acronym: TORICIOL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aurolab (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1PN1011037
Record Dates: First submitted 2011-07-14; First posted 2011-07-19 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2011-07

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): The enrolled subject will be implanted with Toric IOL manufactured by AuroLab
  Interventions: Device: Experimental - Toric Intraocular lenses

INTERVENTIONS:
Device: Experimental - Toric Intraocular lenses — Toric Intraocular Lenses will be implenated with cataract patients having astigmatism

SUMMARY:
The purpose of this study is to measure visual acuity and Intraocular Lens (IOL) rotational stability after implantation of TORIC IOL and to assess the post operative complications after implantation of TORIC IOL.

DETAILED DESCRIPTION:
Among available methods for treating astigmatism in cataract surgery, the implantation of toric IOLs is an emerging technology that shows promising results. Similar to implanting a one-piece acrylic lens, toric IOLs provide good distance vision and, in many patients, freedom from spectacles for distance vision. A low absolute residual refractive cylinder has been associated with the implantation of toric IOLs, and the safety profile for toric IOLs has been good. As improvements with regard to rotational stability and treatment and cylinder power range are made, toric IOLs will emerge as an effective, safe treatment option for correcting astigmatism during cataract surgery.

Further, to evidence on the safety and efficacy of TORIC IOL for patients having cataract associated with astigmatism served as the basis for us to identify the published literature on the safety and efficacy of TORIC IOL implantation in the treatment of cataract associated with astigmatism, thus provide a background for the development of clinical investigation plan for the present study.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 to 65
* Senile cataract
* Posterior Sub Capsular Cataract (PSCC)
* Astigmatism 1.25 D or more
* Residence within 100 kms of Madurai

Exclusion Criteria:

* Traumatic & Complicated cataract
* Poor mydriasis
* Amblyopia
* Severe Pseudo exfoliation (PXF)
* Dense posterior polar cataract (PPC)
* One eyed patients
* Uveitis
* Corneal pathology / Scar
* Retinal Pathology contributing to visual loss
* Intraoperative complication like PC rupture, Zonular dialysis

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-08; Primary Completion 2013-05 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
vision improvement | 150 days
  The visual acuity will be measured after iol implantation on 1 day, 10 days, 40 days and 150 days post operatively

SECONDARY OUTCOMES:
Refractive error correction | 150 days
  To measure the refraction error after IOL implantation on 1 day, 10 days, 40 days and 150 days post operatively

CONTACTS AND LOCATIONS:
Overall Officials: Dr. SHIVKUMAR CHANDRASHEKAR, MBBS., MS.,, Principal Investigator — HOD of IOL & Cataract clinic, Aravind Eye Hospital, Tirunelveli
Locations (1):
- Aravind Eye Hospital, Madurai, Tamil Nadu, India